CLINICAL TRIAL: NCT03751605
Title: Validation of the Respiratory Quotient Measurement Measured Indirectly in Unipulmonary Ventilation (UNIQ Study)
Brief Title: Indirect Measurement of Respiratory Quotient in Unipulmonary Ventilation.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0047
Record Dates: First submitted 2018-11-08; First posted 2018-11-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Respiratory Quotient Measurement
Keywords: unipulmonary ventilation, complications, respiratory quotient.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: unipulmonary ventilation — observational study based on the computation of respiratory quotient in patient cohort treated by unipulmonary ventilation in routine thoracic surgery

SUMMARY:
The measurement of VO2 and VCO2 makes it possible to calculate the respiratory quotient (RQ) (VCO2 / VO2) which is a reflection of human energy metabolism and therefore of anaerobiosis. A study has been conducted in our department to demonstrate the ability of the indirectly measured respiratory quotient (RQ) from the inspired and exhaled breath analysis of the anesthetic respirator to predict the onset of anaerobic metabolism and postoperative complications in the operating room.

Unipulmonary ventilation is the rule in thoracic surgery: it improves surgical exposure and protects the operated lung.

However, no study has examined the impact of these mechanisms on the indirect measurement of RQ in unipulmonary ventilation. The main objective of our work is to validate indirect RQ measurement during unipulmonary ventilation. The secondary objective was to assess the predictability of postoperative complications of indirect QR.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Adults admitted to the operating room for thoracic surgery requiring unipulmonary ventilation

Exclusion Criteria:

* Cardiac surgery
* Laparoscopy
* Preoperative oxygen therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Age>18 years old
  * Adults admitted to the operating room for thoracic surgery requiring unipulmonary ventilation
  Exclusion Criteria:
  * Cardiac surgery
  * Laparoscopy
  * Preoperative oxygen therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Indirect respiratory quotient | during surgery

SECONDARY OUTCOMES:
occurrence of at least one post-operative complication | through study completion, an average of 6 months
  the aim is to predict the occurrence of at least one complication with the use of indirect respiratory quotient

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France